CLINICAL TRIAL: NCT06438432
Title: Trunk Activity Rehabilitation in Young Children With Cerebral Palsy
Acronym: Activ'Tronc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01969-36
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Children With Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RH-RAIT (Experimental): A first group of children will continue their usual rehabilitation (RH) for the first 3 months and then have RAIT for the following 9 months.
  Interventions: Other: RAIT
- RAIT-RAIT (Experimental): The second group of children will have RAIT from the outset during the 12 months of the study.
  Interventions: Other: RAIT

INTERVENTIONS:
Other: RAIT — The RAIT program focuses on improving postural control and balance of the entire body, including the trunk and other affected muscles, through autonomous actions in intermediate postures. This approach uses fundamental automatic control of postural support and balance to enhance the use of affected muscles during all postural and locomotor tasks. The child controls their balance during various voluntary actions from intermediate postures like alternating between four-legged and cobra postures, or swinging from the camel posture. These actions, less difficult than standing and walking, are expected to benefit the latter. The child also performs more challenging trunk movements, requiring dissociation of scapular and pelvic girdle movements or reducing lumbar lordosis.

SUMMARY:
Children with CP exhibit trunk control issues from early childhood, affecting their balance and gait. These issues manifest as unstable walking, increased step width, and more pronounced anterior deceleration of the sternum. Previous studies have shown that early action of the triceps surae compensates for the deficit in trunk postural control. Rehabilitation targeting the trunk has shown significant improvements in postural control and gait.

The main objective is to demonstrate that RAIT (Rehabilitation by Activities Involving the Trunk) significantly reduces the peak anterior deceleration of the sternum at the beginning of the stance phase during barefoot spontaneous walking, with an enhanced effect from prolonged RAIT duration.

Secondary objectives include reducing the downward deceleration of the fifth lumbar vertebra (L5), step width, gait variability index, and improving scores on the early clinical balance scale and the global motor function evaluation.

Participants, children with spastic paraparesis or spastic hemiparesis capable of walking independently, are divided into two groups: one group continuing their usual rehabilitation for 3 months followed by RAIT for 9 months (RH-RAIT), and one group following RAIT for 12 months (RAIT-RAIT). RH involves rehabilitation exercises for lower limb muscles, while RAIT focuses on improving trunk postural control through activities involving intermediate postures.

Functional motor assessments will be conducted initially, then at 3, 6, and 12 months. These include clinical evaluations, gait analysis (step width, gait variability index, anterior foot support), and an analysis of static standing displacement using an inertial sensor placed at L5.

At M0, children with CP are expected to show higher values for deceleration peaks and gait variability indices, and lower scores on evaluation scales compared to typically developing (TD) children. After RAIT, an improvement in judgment criteria is expected: reduction in deceleration peaks, cycle width, gait variability index, anterior foot support, and an increase in scores on the ECPE and EMFG-66-SI.

This study aims to confirm that rehabilitation through trunk-involving activities is more effective than usual rehabilitation in improving postural control and gait dynamics in young children with cerebral palsy, suggesting that this approach could become a standard rehabilitation practice from early childhood.

ELIGIBILITY:
Inclusion Criteria:

For children with CP

* Age between 18 months and 5 years 6 months
* CP type: spastic paraparesis or spastic hemiparesis, GMFCS I to II
* No or moderate retraction of the sural triceps (ankle dorsiflexion: > 5° on clinical examination, knee straight)
* Sufficient level of understanding to carry out activities involving the trunk in the form of self-exercises (rehabilitation protocol), as well as clinical assessments and functional explorations.
* Acceptance by the physiotherapist in charge of the child's follow-up to collaborate in carrying out the RAIT.
* Affiliated with a social security scheme

For children with DT

* Age between 18 months and 5 years 6 months
* Walking acquired before age 18 months
* Sufficient level of understanding to perform clinical assessments and functional explorations
* Affiliated with a social security scheme

Exclusion Criteria:

For children with CP

* Previous surgery on lower limbs less than 1 year ago
* Botulinum toxin A injection less than 6 months ago
* Any change in rehabilitative and/or orthopedic management in the last 2 months
* Hip flessum > 20
* Presence of subacute or chronic pain on standing or walking

For children with DT

- Neurological and/or orthopedic disorders that may influence gait

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Peak anterior deceleration of the sternum at the start of weight-bearing | At inclusion, then 3, 6 and 12 months later
  Varaible obtained via the analysis of walking on a zeno treadmill. A reduced value is expected after RAIT rehabilitation.

SECONDARY OUTCOMES:
EMFG-66-SI | At inclusion, then 3, 6 and 12 months later
  The Evaluation Motrice Fonctionnelle Globale 66 (EMFG-66) is a standardized 66-item clinical score used to assess global motor function and its evolution over time in children with cerebral palsy. The EMFG-66-SI is a faster (approx. 20 to 30 minutes vs. 60 to 80 minutes), validated scoring method for the EMFG-66, using 15 to 39 items. The higher the score, the better.
The Early Clinical Balance Scale | At inclusion, then 3, 6 and 12 months later
  This is a 13-item clinical scale for assessing postural stability (balance ability) in children with cerebral palsy, with two subscales: one dedicated to head and trunk postural control, the other to sitting and standing postural control.The scale has been validated for children aged 1.5 to 11, regardless of GMFCS level (40,47). The scale has been validated for children aged 1.5 to 11, regardless of GMFCS level.)The optimal score is 100. Administering the scale takes around 15 minutes. The higher the score, the better.
Global Motor Function Classification System family report questionnaire | At inclusion
  This questionnaire for parents, based on the child's voluntary movements for sitting, transferring and mobility, provides a 5-level classification of the severity of the child's cerebral palsy. Score between 1 and 5. The higher the score, the more severe the cerebral palsy.
"Reach out" questionnaire | At inclusion, then 3, 6 and 12 months later
  This is a questionnaire designed for parents to assess the upper limb and hand abilities in different functional situations of their child with CP. This questionnaire, validated for children with CP from the age of 2, will help to assess the expected improvement in hand and upper limb function linked to RAIT. The higher the score, the better.
Neuro-orthopaedic assessment | At inclusion, then 3, 6 and 12 months later
  This examination consists of measuring the amplitude of movement of the main joints in one or more planes, using a goniometer. Check against standards for each joint
Neuro-orthopaedic assessment | At inclusion, then 3, 6 and 12 months later
  This examination consists of measuring spasticity of the main muscles, by mobilizing a joint at slow and then fast speed to elicit a stretch reflex. Score between 0 and 4. 4 indicates the highest level of spasticity.
Neuro-orthopaedic assessment | At inclusion, then 3, 6 and 12 months later
  This examination consists of measuring the muscular strength of the main muscle groups, by asking the subject to mobilize a joint against resistance. Score between 0 and 5. The higher the score, the better.
peak downward deceleration of L5 at the start of support | At inclusion, then 3, 6 and 12 months later
  varaible obtained via the analysis of walking on a zeno treadmill. A reduced value is expected after RAIT rehabilitation.
Gait variability index | At inclusion, then 3, 6 and 12 months later
  Composite score based on 9 spatio-temporal parameters that quantifies the distance between the amount of variability observed in an asymptomatic reference group and the amount of variability observed in the patient. This index assesses gait instability and the risk of falling. It is usually high in children with CP.
Cycle width | At inclusion, then 3, 6 and 12 months later
  Varaible obtained via the analysis of walking on a zeno treadmill. A reduced value is expected after RAIT rehabilitation.
Anterior support of the foot during 1st double support | At inclusion, then 3, 6 and 12 months later
  Ratio between the integrated pressure of the forefoot and the integrated pressure of the whole foot during the 1st double support. This variable will be higher the more the foot is supported on the ground by the forefoot, as in the PC child, and lower the more the foot is supported by the heel, as in the typically developing child.
Edinburgh walk visual score | At inclusion, then 3, 6 and 12 months later
  Score developed for children with cerebral palsy, assessing the extent of kinematic deviations compared to typically developing children. (0 = normal, 1 = moderate or mild pathology, 2 = severe pathology). So 0 here means the best EVGS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France

IPD SHARING:
Plan to Share IPD: No